CLINICAL TRIAL: NCT06432608
Title: Single Arm Study to Evaluate the Efficacy of Lacticaseibacillus Paracasei Strain Shirota (Formerly Lactobacillus Casei Strain Shirota) Fermented Milk (Yakult®) on the Maintenance of Clinical Manifestations of Functional Constipation in Mexican Adults
Brief Title: Efficacy of Lacticaseibacillus Paracasei Strain Shirota on Clinical Manifestation of Functional Constipation in Mexican Adults
Acronym: FC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guadalajara (Other)
Collaborators: Yakult Honsha Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UDG-FC-2024
Record Dates: First submitted 2024-05-09; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Constipation
Keywords: functional constipation; clinical manifestation; mexican; short fatty acids; Lacticaseibacillus paracasei strain Shirota
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: Original longitudinal, analytical, and prospective quasi-experimental study in adults diagnosed with functional chronic constipation under the ROME IV criteria. The study will provide a product based on fermented milk with the probiotic Lacticaseibacillus paracasei strain Shirota for 4 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): The single arm contemplates providing the study subjects diagnosed with functional constipation with a product based on fermented milk (80mL) daily for 4 weeks.
  Interventions: Dietary Supplement: fermented milk, Yakult

INTERVENTIONS:
Dietary Supplement: fermented milk, Yakult — Study subjects will be provided with a product based on fermented milk, Yakult (80mL) daily for four weeks in order to know the effects of clinical manifestation of functional constipation and short-fatty acids in the Mexican population

SUMMARY:
Chronic functional constipation is a gastrointestinal disorder with an approximate prevalence of 14% of the Mexican population, which is characterized by difficult or incomplete defecation and/or infrequent bowel movements, with the absence of symptoms such as abdominal pain or inflammation, and in If they occur, they should not be the predominant symptoms. Its origin is multifactorial and includes variables such as diet, water consumption, alteration in motility, and intestinal microbiota, the latter as a source of different secondary metabolites such as short-chain fatty acids (SCFAs).

Lower SCFA values in constipation would alter the relationship between them, increasing the risk of clinical manifestations of functional chronic constipation. In addition to physical discomfort, subjects with this disease manifest alterations in their quality of life.

Recent studies have suggested using probiotic microorganisms to treat this functional disorder due to their beneficial effects on evacuation frequency, SCFAs, and quality of life. However, in Mexico, knowledge of the above is limited. Therefore, this research aims to determine the effect of consuming a product based on fermented milk with the probiotic Lacticaseibacillus paracasei strain Shirota on the clinical manifestations of functional constipation in Mexican adults and its relationship with SCFAs.

DETAILED DESCRIPTION:
1. Background

   Constipation is an intestinal disorder characterized by difficulty defecating, infrequent bowel movements, hard or lumpy stools, excessive straining, a feeling of incomplete evacuation, and, in some cases, the use of manual techniques to facilitate evacuation.

   Due to its presentation time, constipation is classified as acute or chronic. The acute one lasts less than a week and is commonly determined by a change in diet and/or lifestyle (low fiber intake, decreased physical activity, stress, going to the bathroom in an unknown place, etc.). For its part, the symptoms of chronic illness have occurred over three to six months. Chronic constipation is among the most common gastrointestinal conditions, usually primary or secondary. The first is a consequence of multiple pathophysiological alterations, such as alteration of colonic regulation, lack of coordination of the neuromuscular apparatus, and dysfunction of the brain-gut axis. In turn, secondary chronic constipation can be caused by drugs, neurological disorders, anatomical processes, or metabolic diseases.

   Chronic constipation is defined "from a clinical point of view, chronic constipation is considered secondary when it is a consequence of metabolic, neurological alterations, structural lesions or medications. When other causes have been excluded, it is considered primary, idiopathic, or functional constipation" (FD).

   1.1. Clinical manifestations

   Chronic constipation is a functional gastrointestinal disorder with a prevalence of 3 to 27%, mainly among women and older adults. Approximately 1 in 6 individuals experience chronic constipation. The Mexican Consensus on chronic constipation mentions a prevalence of 14.4% in Mexicans, while other studies carried out in the country have reported a prevalence between 2.4 and 22.3%.

   This pathology is considered a syndrome with different symptoms that are expressed variably. For this reason, the ROMA (Rome Foundation for Functional Gastrointestinal Problems) criteria have been used to diagnose functional chronic constipation. In 2016, the ROMA criteria updated their guidelines, currently in version IV, and included eight categories: A) esophageal disorders; B) gastroduodenal disorders; C) intestinal disorders; D) gastrointestinal pain of centrally median disorders; E) disorders of the sphincter of Oddi and the gallbladder; F) anorectal disorders; G) functional gastrointestinal disorders of childhood and G) functional gastrointestinal disorders of adolescence. Functional intestinal disorders are defined by these criteria, which allow us to differentiate the symptoms of patients with chronic functional constipation from those with similar clinical conditions, such as irritable bowel syndrome.

   In the ROME IV criteria, chronic functional constipation is a disorder characterized by persistent or incomplete difficult defecation and/or infrequent bowel movements without symptoms such as abdominal pain and/or inflammation or, if present, that are not the predominant symptoms. The Bristol scale supports the criteria in which grades 1 and 2 correspond to constipation and correlate with prolonged intestinal transit.

   1.2. Constipation and short-chain fatty acids

   Chronic constipation is a multifactorial process influenced by diet, stool volume, water content, and intestinal microbiota. In recent years, it has been considered that alterations in the balance of the intestinal microbiota may influence the clinical manifestations of chronic constipation. It has been reported that the intestinal microbiota of constipated patients differs from that of healthy adults and children, with a decrease in the genera Lactobacillus and Bifidobacterium. Studies with gnotobiotic animals and in vitro have suggested that the intestinal microbiota influences intestinal motility, the integrity of the intestinal barrier, the modulation of colonic pH, and the immune or nervous response through the production of short-chain fatty acids: butyrate, propionate, and acetate.

   1.3. Constipation and probiotics

   Patients with constipation usually have a prolonged intestinal transit time compared to healthy subjects, decreasing evacuation frequency and stool consistency. To achieve this, laxatives, dietary fiber supplements, and the prescription of some drugs are used as treatment. However, in recent years, the use of probiotics has been considered due to the impact of their consumption on the intestinal microbiota/metabolites and, in turn, on gastric motility.

   It has been reported that consuming 10^8 to 3 x 10^10 CFU per day of specific probiotic strains improves intestinal transit, increases evacuation frequency, and improves symptoms related to constipation. Studies with Lacticaseibacillus paracasei strain Shirota (LcS) in the Chinese population showed improvement in the frequency and consistency of fecal matter and reduced intestinal discomfort. The intake of probiotics improves intestinal transit and increases the levels of organic acids that promote peristalsis. It also increases the Bifidobacterium and Lactobacillus genera, which are usually in lower abundance in constipation. Probiotics could not only directly improve intestinal discomfort but also through the formation of secondary metabolites of the intestinal microbiota, such as short-chain fatty acids.

   Therefore, probiotics such as Lacticaseibacillus paracasei strain Shirota have begun to be studied in murine models and in the Asian population as a non-pharmacological alternative for functional chronic constipation. However, its effect on the Mexican population with constipation requires more evidence, as does the relationship between the intake of probiotics in functional constipation and short-chain fatty acids.
2. General objective:

   To evaluate the efficiency of Lacticaseibacillus paracasei strain Shirota Shirota (formerly Lactobacillus casei strain Shirota) in fermented milk (Yakult®) on the maintenance of the clinical manifestations of functional constipation in Mexican adults.
3. Hypothesis:

   The consumption of a product based on milk fermented with Lacticaseibacillus paracasei strain Shirota, has an effect on the maintenance of the clinical manifestations of functional constipation in Mexican adults.
4. Methodology:

An original longitudinal, analytical, and prospective quasi-experimental study in adults diagnosed with functional chronic constipation under the ROME IV criteria is planned. The study will provide a product based on fermented milk with the probiotic Lacticaseibacillus paracasei strain Shirota for four weeks. Before consuming the product, a baseline analysis of SCFAs will be carried out in fecal matter. As part of the techniques and procedures, height and weight will be measured using the ISAK methodology to obtain the body mass index (BMI). Meanwhile, the clinical manifestations of evacuation frequency and consistency of fecal matter will be evaluated, considering the ROME IV criteria, with visual support from the Bristol and symptom severity scales. The analysis of short-chain fatty acids will be done by gas chromatography, whose signal will be compared with an internal standard.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 20 and 60 years old, diagnosed with functional chronic constipation (according to the Rome IV criteria).
* Men and women who have given informed consent.

Exclusion Criteria:

* Constipation due to neurological, pharmacological or organic causes.
* Pregnancy or pregnancy expected within the next month.
* Breastfeeding women.
* Diagnosed pathologies such as: diabetes mellitus, kidney or liver failure, infectious disease, inflammatory disease or any neoplastic disease.
* Use of laxatives within 14 days prior to the start of the intervention.
* Use of antibiotics within 14 days prior to the start of the intervention.
* Diagnosis of cancer in the last three years.
* History of drug and medication abuse.
* Active alcoholism with a daily intake greater than 50 g/day.
* Lactose intolerance.
* Known allergies to any substance in the study product (e.g., cow's milk proteins).
* Any subject who needs manual maneuvers to evacuate feces.
* Anticipated major changes in diet or exercise during the study period.
* Eating disorders.
* Participation in another study with any investigational product within 3 months prior to enrollment.
* Regular Yakult consumers
* Subject who does not have the capacity to consent.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-11-25 (Estimated); Study Completion 2025-11-25 (Estimated)

PRIMARY OUTCOMES:
Clinical manifestation of functional constipation | 2 months
  Clinical manifestation will be measure by Bristol scale (1-2 hard stools; 3-4 normal; 4-5 soft stools), Frequency of bowel movements will be obtained by the question of how many times per week have defecated, meanwhile severity of symptoms related to constipation will include indicators of difficulty passing stool, pain, and feeling of incomplete evacuation on a 4-point scale (1, none; 2, a little; 3, some; and 4, a lot)

SECONDARY OUTCOMES:
Analysis of short-chain fatty acids | 2 months
  The short chain fatty acids acetate, butyrate and propionate will be analyzed from the fecal material sample. Fatty acids will be measured by gas chromatography equipped with a flame ionization detector and a MEGA-ACID (FFAD) chromatographic column of 30.0m length, with internal diameter: 0.25 ID, thickness: 0.40 µm and 3µL injector. Samples will be analyzed by chromatographic method through the MEGA-ACID column, with an injection of 3 µL and whose injection mode is Split 1:25. The column flow will be 3.0 mL/min, in 29 min at 250°C, with a gas flow of N2 30.0mL/min, H2 40mL/min, Air 400 mL/min. The signal ratio (peak area ratio) of the short chain fatty acid compared to internal standards: acetic acid (71251 Sigma-Aldrich), propionic acid (94425 Sigma-Aldrich), butyric acid (19215 Sigma-Aldrich); in a range of 3.13-400ppm. It will later be corrected by the relative correction factor. The above will be used to calculate the concentration of the short chain fatty acid.
Height | 2 months
  Height (mt) it will be recorded which technique extension requires the subject to stand with the feet apart at a 45° angle and the heels together, the posterior aspect of the buttocks and the upper back resting on the stadiometer.The head should be in the Frankfort plane. The subject is asked to take a deep breath and hold it, The scorer places the square triangular piece firmly over the vertex, squeezing the hair as tightly as possible. The measurement is taken at the end of a deep breath.
Body weight | 2 months
  Body weight (kg) will be checked that the scale is in the zero register. Then the subject stands in the center of it without support and with the weight distributed evenly between both feet. The head should be elevated and the eyes looking directly forward.
Body Mass Index (BMI) | 2 months
  The body mass index (BMI) will be calculated by dividing the weight, previously obtained from the person evaluated, by the squared height (mt). BMI will be reported in categories: <18.5, 18.5 - 24.9, 25-29.9 and >30

CONTACTS AND LOCATIONS:
Overall Officials: Ma.Refugio Torres Vitela, PhD, Principal Investigator — University of Guadalajara

IPD SHARING:
Plan to Share IPD: No
This is a project that involves data about patent

REFERENCES:
- [Background] Aziz I, Whitehead WE, Palsson OS, Tornblom H, Simren M. An approach to the diagnosis and management of Rome IV functional disorders of chronic constipation. Expert Rev Gastroenterol Hepatol. 2020 Jan;14(1):39-46. doi: 10.1080/17474124.2020.1708718. Epub 2020 Jan 2. PMID 31893959
- [Background] Araujo MM, Botelho PB. Probiotics, prebiotics, and synbiotics in chronic constipation: Outstanding aspects to be considered for the current evidence. Front Nutr. 2022 Dec 8;9:935830. doi: 10.3389/fnut.2022.935830. eCollection 2022. PMID 36570175
- [Background] Chen S, Ou Y, Zhao L, Li Y, Qiao Z, Hao Y, Ren F. Differential Effects of Lactobacillus casei Strain Shirota on Patients With Constipation Regarding Stool Consistency in China. J Neurogastroenterol Motil. 2019 Jan 31;25(1):148-158. doi: 10.5056/jnm17085. PMID 30646486
- [Background] Cheng Y, Liu J, Ling Z. Short-chain fatty acids-producing probiotics: A novel source of psychobiotics. Crit Rev Food Sci Nutr. 2022;62(28):7929-7959. doi: 10.1080/10408398.2021.1920884. Epub 2021 May 6. PMID 33955288
- [Background] Dimidi E, Christodoulides S, Fragkos KC, Scott SM, Whelan K. The effect of probiotics on functional constipation in adults: a systematic review and meta-analysis of randomized controlled trials. Am J Clin Nutr. 2014 Oct;100(4):1075-84. doi: 10.3945/ajcn.114.089151. Epub 2014 Aug 6. PMID 25099542
- [Background] Forootan M, Bagheri N, Darvishi M. Chronic constipation: A review of literature. Medicine (Baltimore). 2018 May;97(20):e10631. doi: 10.1097/MD.0000000000010631. PMID 29768326
- [Background] Lange O, Proczko-Stepaniak M, Mika A. Short-Chain Fatty Acids-A Product of the Microbiome and Its Participation in Two-Way Communication on the Microbiome-Host Mammal Line. Curr Obes Rep. 2023 Jun;12(2):108-126. doi: 10.1007/s13679-023-00503-6. Epub 2023 May 19. PMID 37208544
- [Background] Markowiak-Kopec P, Slizewska K. The Effect of Probiotics on the Production of Short-Chain Fatty Acids by Human Intestinal Microbiome. Nutrients. 2020 Apr 16;12(4):1107. doi: 10.3390/nu12041107. PMID 32316181
- [Background] Morrison DJ, Preston T. Formation of short chain fatty acids by the gut microbiota and their impact on human metabolism. Gut Microbes. 2016 May 3;7(3):189-200. doi: 10.1080/19490976.2015.1134082. Epub 2016 Mar 10. PMID 26963409
- [Background] Simren M, Palsson OS, Whitehead WE. Update on Rome IV Criteria for Colorectal Disorders: Implications for Clinical Practice. Curr Gastroenterol Rep. 2017 Apr;19(4):15. doi: 10.1007/s11894-017-0554-0. PMID 28374308
- [Background] Schmulson Wasserman M, Francisconi C, Olden K, Aguilar Paiz L, Bustos-Fernandez L, Cohen H, Passos MC, Gonzalez-Martinez MA, Iade B, Iantorno G, Ledesma Ginatta C, Lopez-Colombo A, Perez CL, Madrid-Silva AM, Quilici F, Quintero Samudio I, Rodriguez Varon A, Suazo J, Valenzuela J, Zolezzi A. [The Latin-American Consensus on Chronic Constipation]. Gastroenterol Hepatol. 2008 Feb;31(2):59-74. doi: 10.1157/13116072. Spanish. PMID 18279643
- [Background] Yuan F, Tan W, Ren H, Yan L, Wang Y, Luo H. The Effects of Short-Chain Fatty Acids on Rat Colonic Hypermotility Induced by Water Avoidance Stress. Drug Des Devel Ther. 2020 Nov 2;14:4671-4684. doi: 10.2147/DDDT.S246619. eCollection 2020. PMID 33173277
- [Background] Zhuang M, Shang W, Ma Q, Strappe P, Zhou Z. Abundance of Probiotics and Butyrate-Production Microbiome Manages Constipation via Short-Chain Fatty Acids Production and Hormones Secretion. Mol Nutr Food Res. 2019 Dec;63(23):e1801187. doi: 10.1002/mnfr.201801187. Epub 2019 Oct 22. PMID 31556210